CLINICAL TRIAL: NCT05089448
Title: Morning Versus Bedtime Dosing of Antihypertensive Medication in Grade 1 Day-night Hypertension: a Multicenter Randomized Controlled Trial (Dosing-Time Trial)
Brief Title: Morning Versus Bedtime Dosing of Antihypertensive Medication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yan Li (Other)
Responsible Party: Sponsor-Investigator, Yan Li, Professor of Cardiovascular Medicine, Shanghai Institute of Hypertension
Organization: Shanghai Institute of Hypertension (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dosing-Time Trial20210118
Record Dates: First submitted 2021-09-27; First posted 2021-10-22 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Blood Pressure; Drug Use
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The morning dosing group (Active Comparator): After randomization, subjects will take alisartan 120 mg (Salubris, Shenzhen, China) once daily at 6:00-10:00. After 8 weeks of treatment, if the 24-hour ambulatory systolic BP remained ≥ 130 mmHg, alisartan will be doubled to 240mg. After 16 weeks of treatment, if the 24-hour ambulatory systolic BP remained ≥ 130 mmHg, amlodipine besylate 2.5 mg (Dawnrays, Suzhou, China) once daily will be added. The whole treatment duration will last for 24 weeks.
  Interventions: Drug: Alisartan, Amlodipine besylate
- The bedtime dosing group (Experimental): After randomization, subjects will take alisartan 120 mg once daily at 20:00-24:00. The follow-up plan is the same as the morning dosing group.
  Interventions: Drug: Alisartan, Amlodipine besylate

INTERVENTIONS:
Drug: Alisartan, Amlodipine besylate — Drugs will be taken once daily at 6:00-10:00.
  Arms: The morning dosing group
Drug: Alisartan, Amlodipine besylate — Drugs will be taken once daily at 20:00-24:00.
  Arms: The bedtime dosing group

SUMMARY:
Previous studies have shown that elevated nighttime blood pressure (BP) was more closely associated with cardiovascular mortality and morbidity than daytime and clinic BPs. With increasingly advanced technology, not only 24-hour ambulatory but also home BP monitors can be used to evaluate nighttime BP. The validation study of the Omron HEM 9601T showed that the wrist-type home BP monitor could be a suitable and reliable tool for the diagnosis and management of nocturnal hypertension. However, up to now, there is no data on home nighttime BP in Chinese patients and it is unclear if different dosing time would reduce ambulatory and home nighttime BPs differently.

The investigators therefore designed a multicenter randomized clinical trial to compare between morning dosing and bedtime dosing of antihypertensive medications in the difference in nighttime, daytime and the 24-h BP reductions evaluated by both ambulatory and home BP monitoring, and in target organ protections.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-70 years old;
2. Never treated for hypertension or stopped using antihypertensive drugs for at least 2 weeks;
3. In the two screenings,the clinical systolic BP should be in the range of 140-159 mmHg, the diastolic BP < 100 mmHg;
4. The average 24-hour systolic BP ≥130mmHg, daytime systolic BP ≥ 135 mmHg, and nighttime systolic BP ≥ 120 mmHg;
5. The average of bilateral brachial-ankle pulse wave velocity ≥14m/s;
6. Be willing to participate in the trial, sign the informed consent form, and be able to visit doctors by himself or herself.

Exclusion Criteria:

1. Secondary hypertension;
2. Concomitant obstructive sleep apnea (STOP-BANG score ≥ 5), insomnia, Parkinson's syndrome, or nocturnal polyuria and other diseases that affect nighttime BP;
3. Need to work at night;
4. Ambulatory BP monitoring was invalid (<70% valid readings, or <20 daytime readings or <7 nighttime readings);
5. Concomitant diseases that need taking medications influencing BP;
6. Coronary heart disease, myocardial infarction or stroke within recent 6 months;
7. Atrial fibrillation or frequent arrhythmia;
8. Abnormal liver function exemplified as an increased alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin (TBL) over the double of the upper limit of normal range; abnormal renal function exemplified as a serum creatinine ≥176 µmol/L; and plasma potassium ≥5.5 mmol/L or ≤3.5mmol/L;
9. Pregnant or lactating women;
10. Contraindications of angiotensin II receptor blocker or calcium channel blocker;
11. Other concomitant diseases which are considered not suitable to participate in the trial, such as thyroid diseases, acute infectious diseases, chronic mental diseases, tumor, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Nighttime systolic BP reduction in mmHg | 24 weeks
  The difference between the morning and bedtime dosing groups in nighttime systolic BP reduction in mmHg measured by the ambulatory BP monitoring after the treatment for 24 weeks

SECONDARY OUTCOMES:
Daytime systolic BP reduction in mmHg, 24-Hour systolic BP reduction in mmHg, Home systolic BP reduction in mmHg | 24 weeks
  The difference between the morning and bedtime dosing groups in the daytime and 24-hour systolic BPs reduction in mmHg measured by the ambulatory BP monitoring and home systolic BP reduction in mmHg after treatment for 24 weeks
Brachial-ankle pulse wave velocity reduction in cm per second | 12 and 24 weeks
  The difference between the morning and bedtime dosing groups in reduction of brachial-ankle pulse wave velocity after treatment for 12 and 24 weeks
Ambulatory night-to-day BP ratio change in percent; proportions of non-dippers in percent, morning systolic blood pressure in mmHg, | 8 weeks and 24 weeks
  The difference between the morning and bedtime dosing groups in change of Ambulatory night-to-day BP ratio change in percent; proportions of non-dippers in percent, and morning systolic blood pressure in mmHg after treatment for 8 and 24 weeks.
Urinary albumine-to-creatinine ratio change in mg/mmol | 12 weeks and 24 weeks
  The difference between the morning and bedtime dosing groups in change of microalbumine-to-creatinine ratio in random urine samples after treatment for 12 weeks and 24 weeks
change in prevalence of left ventricular hypertrophy defined based on electrocardiogram | 12 weeks and 24 weeks
  The difference between the morning and bedtime dosing groups in the change in prevalence (percentage) of left ventricular hypertrophy defined based on Cornell product and Sokolow-Lyon index in electrocardiogram after treatment for 12 weeks and 24 weeks
change in prevalence of left ventricular hypertrophy defined based on echocardiography | 24 weeks
  prevalence (percentage) of left ventricular hypertrophy defined based on left ventricular mass index assessed by echocardiography after treatment for 24 weeks
Serum uric acid in umol/L | 24 weeks
  The difference between the morning and bedtime dosing groups in serum uric acid in umol/L after treatment for 24 weeks
The difference in daytime systolic and diastolic BPs between the ambulatory and home BP monitoring at baseline and after treatment for 24 weeks | 24 weeks
  The difference in daytime systolic and diastolic BPs between the ambulatory and home BP monitoring at baseline and after treatment for 24 weeks
The difference in nighttime systolic and diastolic BPs between the ambulatory and home BP monitoring at baseline and after treatment for 24 weeks | 24 weeks
  The difference in nighttime systolic and diastolic BPs between the ambulatory and home BP monitoring at baseline and after treatment for 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China